CLINICAL TRIAL: NCT00722878
Title: Early Onset and Progression of Primary Ciliary Dyskinesia Lung Disease Prior to 10 Years of Age
Brief Title: Long-term Lung Function and Disease Progression in Children With Early Onset Primary Ciliary Dyskinesia Lung Disease
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-0764; U54HL096458 (NIH); RDCRN 5903 (Other: UNC)
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Kartagener Syndrome
Keywords: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Kartagener Syndrome; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 2 teaspoons of blood and a small amount of urine (if the child is able to urinate in a cup) will be collected and held at the specimen bank located at Denver Children's Hospital. These samples will be used to help identify markers that may predict the clinical course of PCD.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary ciliary dyskinesia (PCD), also known as Kartagener syndrome, is a genetic disorder of the cilia, which are microscopic hair-like cells. Cilia work to keep the respiratory system clean by moving mucus that contains debris to the large airways, where it can be coughed out. People with PCD have cilia that do not move properly and therefore are not effective in cleaning the respiratory system. This study will determine when PCD starts and how it changes over time, specifically in terms of how well the lungs work, what germs grow in lung secretions, and how the lungs look on computed tomography (CT) scans.

DETAILED DESCRIPTION:
PCD, or Kartagener syndrome, is a genetic disorder that causes hair-like cells called cilia to move improperly, or in some cases, not at all. Cilia are needed to help clear the respiratory system of pollutants. When they work properly, they move debris-filled mucus into the large airways, allowing the debris to be coughed out of the body. When the cilia do not work properly, the body cannot rid itself of debris and is left vulnerable to serious infections in the sinuses, ears, and lungs. Over time, repeated infections can lead to scarring and permanent obstruction of these body areas. This study will determine when PCD starts and how it changes over time, specifically in terms of how well the lungs work, what germs grow in lung secretions, and how the lungs look on CT scans. This research may lead to a better understanding of PCD and thereby help doctors improve clinical management of the disease.

Children in this study will attend six study visits over 5 years. At the first visit, parents will review their child's medical and cough history with doctors. Also at this visit, children will undergo a physical exam that will include measures of temperature, blood pressure, heart rate, respiration rate, and oxygen saturation level. Additional procedures will include collection of a respiratory mucus sample or a throat culture, measurement of nasal nitric oxide, collection of blood and urine for specimen banking, a CT scan, and lung function testing. Children younger than 3 years of age will undergo the scan and lung function test under sedation. Children older than 3 years of age will not receive sedation. CT scans will be performed at the initial visit and during the visits 3 and 5 for children older than 3. For children younger than 3 years, chest CT scans will be performed at the initial visit and during visits 4 and 6. Lung function tests and blood and urine collection may be repeated at some of the remaining yearly visits. Between yearly visits, parents will track on a calendar their children's use of oral, inhaled, and intravenous antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 5 years of age
* Diagnosis of PCD or probable PCD based on criteria listed above
* Parent or legal guardian willing to give informed consent

Exclusion Criteria:

* Unable to attend follow-up appointments
* History of lung transplant
* Any co-existing severe diseases that may have significant impact on lung function, respiratory infections, or overall health status (i.e., severe congenital heart disease, severe scoliosis, AIDS, cancer, or end-stage kidney disease)

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants in this study will be children younger than 5 years of age who have been diagnosed with PCD as based on electron microscopy and/or presence of two known disease-causing gene mutations or for whom a diagnosis of PCD has been determined probable as based on clinical features and very low nasal nitric oxide (less than 60 nl/minute).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-07; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Infant lung function | Measured at initial study visit (for children under 3)
Spirometry measures | Measured yearly for 5 years (after age of 3 years)
Respiratory cultures | Measured yearly for 5 years
Chest CT scan results | Measured at the initial study visit and at Years 3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Margaret W. Leigh, MD, Study Chair — University of North Carolina, Chapel Hill; Margaret Rosenfeld, MD, MPH, Study Chair — Seattle Children's Hospital; Stephanie Davis, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (6):
- United States (5):
  - Stanford University, Palo Alto, Palo Alto, California
  - The Children's Hospital, Denver, Denver, Colorado
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital and Regional Medical Center, Seattle, Seattle, Washington
- The Hospital for Sick Children, Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Imbrie JD. Kartagener's syndrome: a genetic defect affecting the function of cilia. Am J Otolaryngol. 1981 Aug;2(3):215-22. doi: 10.1016/s0196-0709(81)80018-x. PMID 6974512
- [Background] Ramotowski R, Guz W, Zieba E, Zlomaniec G. Clinical and radiological aspects of Kartagener's syndrome. Ann Univ Mariae Curie Sklodowska Med. 2001;56:151-5. PMID 11977302
- [Background] Newmark H 3rd, Willis G, Ablemayor E, Chakmakian V. Kartagener's syndrome seen on CT. Comput Radiol. 1985 Sep-Oct;9(5):279-81. doi: 10.1016/0730-4862(85)90052-6. PMID 3877608
- [Background] Griggs RC, Batshaw M, Dunkle M, Gopal-Srivastava R, Kaye E, Krischer J, Nguyen T, Paulus K, Merkel PA; Rare Diseases Clinical Research Network. Clinical research for rare disease: opportunities, challenges, and solutions. Mol Genet Metab. 2009 Jan;96(1):20-6. doi: 10.1016/j.ymgme.2008.10.003. Epub 2008 Nov 13. PMID 19013090
- [Background] Lie H, Zariwala MA, Helms C, Bowcock AM, Carson JL, Brown DE 3rd, Hazucha MJ, Forsen J, Molter D, Knowles MR, Leigh MW, Ferkol TW. Primary ciliary dyskinesia in Amish communities. J Pediatr. 2010 Jun;156(6):1023-1025. doi: 10.1016/j.jpeds.2010.01.054. Epub 2010 Mar 29. PMID 20350728
- [Background] Olin JT, Burns K, Carson JL, Metjian H, Atkinson JJ, Davis SD, Dell SD, Ferkol TW, Milla CE, Olivier KN, Rosenfeld M, Baker B, Leigh MW, Knowles MR, Sagel SD; Genetic Disorders of Mucociliary Clearance Consortium. Diagnostic yield of nasal scrape biopsies in primary ciliary dyskinesia: a multicenter experience. Pediatr Pulmonol. 2011 May;46(5):483-8. doi: 10.1002/ppul.21402. Epub 2011 Jan 31. PMID 21284095
- [Background] Zariwala MA, Omran H, Ferkol TW. The emerging genetics of primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):430-3. doi: 10.1513/pats.201103-023SD. PMID 21926394
- [Background] Leigh MW, O'Callaghan C, Knowles MR. The challenges of diagnosing primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):434-7. doi: 10.1513/pats.201103-028SD. PMID 21926395
- [Background] Sagel SD, Davis SD, Campisi P, Dell SD. Update of respiratory tract disease in children with primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):438-43. doi: 10.1513/pats.201103-024SD. PMID 21926396
- [Background] Davis SD, Knowles M, Leigh M. Introduction: primary ciliary dyskinesia and overlapping syndromes. Proc Am Thorac Soc. 2011 Sep;8(5):421-2. doi: 10.1513/pats.201103-026SD. No abstract available. PMID 21926392
- [Background] Ostrowski LE, Dutcher SK, Lo CW. Cilia and models for studying structure and function. Proc Am Thorac Soc. 2011 Sep;8(5):423-9. doi: 10.1513/pats.201103-027SD. PMID 21926393
- [Background] Mateos-Corral D, Coombs R, Grasemann H, Ratjen F, Dell SD. Diagnostic value of nasal nitric oxide measured with non-velum closure techniques for children with primary ciliary dyskinesia. J Pediatr. 2011 Sep;159(3):420-4. doi: 10.1016/j.jpeds.2011.03.007. Epub 2011 Apr 22. PMID 21514598
- [Background] Knowles MR, Leigh MW, Carson JL, Davis SD, Dell SD, Ferkol TW, Olivier KN, Sagel SD, Rosenfeld M, Burns KA, Minnix SL, Armstrong MC, Lori A, Hazucha MJ, Loges NT, Olbrich H, Becker-Heck A, Schmidts M, Werner C, Omran H, Zariwala MA; Genetic Disorders of Mucociliary Clearance Consortium. Mutations of DNAH11 in patients with primary ciliary dyskinesia with normal ciliary ultrastructure. Thorax. 2012 May;67(5):433-41. doi: 10.1136/thoraxjnl-2011-200301. Epub 2011 Dec 18. PMID 22184204
- [Background] Stillwell PC, Wartchow EP, Sagel SD. Primary Ciliary Dyskinesia in Children: A Review for Pediatricians, Allergists, and Pediatric Pulmonologists. Pediatr Allergy Immunol Pulmonol. 2011 Dec;24(4):191-196. doi: 10.1089/ped.2011.0099. PMID 22276227
- [Background] Knowles MR, Leigh MW, Zariwala MA. Cutting edge genetic studies in primary ciliary dyskinesia. Thorax. 2012 May;67(5):464; author reply 464. doi: 10.1136/thoraxjnl-2012-201609. Epub 2012 Feb 10. No abstract available. PMID 22328589
- [Background] Horani A, Druley TE, Zariwala MA, Patel AC, Levinson BT, Van Arendonk LG, Thornton KC, Giacalone JC, Albee AJ, Wilson KS, Turner EH, Nickerson DA, Shendure J, Bayly PV, Leigh MW, Knowles MR, Brody SL, Dutcher SK, Ferkol TW. Whole-exome capture and sequencing identifies HEATR2 mutation as a cause of primary ciliary dyskinesia. Am J Hum Genet. 2012 Oct 5;91(4):685-93. doi: 10.1016/j.ajhg.2012.08.022. PMID 23040496
- [Background] Ferkol TW, Leigh MW. Ciliopathies: the central role of cilia in a spectrum of pediatric disorders. J Pediatr. 2012 Mar;160(3):366-71. doi: 10.1016/j.jpeds.2011.11.024. Epub 2011 Dec 16. No abstract available. PMID 22177992
- [Background] Nakhleh N, Francis R, Giese RA, Tian X, Li Y, Zariwala MA, Yagi H, Khalifa O, Kureshi S, Chatterjee B, Sabol SL, Swisher M, Connelly PS, Daniels MP, Srinivasan A, Kuehl K, Kravitz N, Burns K, Sami I, Omran H, Barmada M, Olivier K, Chawla KK, Leigh M, Jonas R, Knowles M, Leatherbury L, Lo CW. High prevalence of respiratory ciliary dysfunction in congenital heart disease patients with heterotaxy. Circulation. 2012 May 8;125(18):2232-42. doi: 10.1161/CIRCULATIONAHA.111.079780. Epub 2012 Apr 12. PMID 22499950
- [Background] Antony D, Becker-Heck A, Zariwala MA, Schmidts M, Onoufriadis A, Forouhan M, Wilson R, Taylor-Cox T, Dewar A, Jackson C, Goggin P, Loges NT, Olbrich H, Jaspers M, Jorissen M, Leigh MW, Wolf WE, Daniels ML, Noone PG, Ferkol TW, Sagel SD, Rosenfeld M, Rutman A, Dixit A, O'Callaghan C, Lucas JS, Hogg C, Scambler PJ, Emes RD; Uk10k; Chung EM, Shoemark A, Knowles MR, Omran H, Mitchison HM. Mutations in CCDC39 and CCDC40 are the major cause of primary ciliary dyskinesia with axonemal disorganization and absent inner dynein arms. Hum Mutat. 2013 Mar;34(3):462-72. doi: 10.1002/humu.22261. Epub 2013 Feb 11. PMID 23255504
- [Background] Sears PR, Thompson K, Knowles MR, Davis CW. Human airway ciliary dynamics. Am J Physiol Lung Cell Mol Physiol. 2013 Feb 1;304(3):L170-83. doi: 10.1152/ajplung.00105.2012. Epub 2012 Nov 9. PMID 23144323
- [Background] Knowles MR, Leigh MW, Ostrowski LE, Huang L, Carson JL, Hazucha MJ, Yin W, Berg JS, Davis SD, Dell SD, Ferkol TW, Rosenfeld M, Sagel SD, Milla CE, Olivier KN, Turner EH, Lewis AP, Bamshad MJ, Nickerson DA, Shendure J, Zariwala MA; Genetic Disorders of Mucociliary Clearance Consortium. Exome sequencing identifies mutations in CCDC114 as a cause of primary ciliary dyskinesia. Am J Hum Genet. 2013 Jan 10;92(1):99-106. doi: 10.1016/j.ajhg.2012.11.003. Epub 2012 Dec 20. PMID 23261302
- [Background] Ferkol TW, Puffenberger EG, Lie H, Helms C, Strauss KA, Bowcock A, Carson JL, Hazucha M, Morton DH, Patel AC, Leigh MW, Knowles MR, Zariwala MA. Primary ciliary dyskinesia-causing mutations in Amish and Mennonite communities. J Pediatr. 2013 Aug;163(2):383-7. doi: 10.1016/j.jpeds.2013.01.061. Epub 2013 Mar 7. PMID 23477994